CLINICAL TRIAL: NCT01481545
Title: Bevacizumab With Pelvic Radiotherapy And Primary Chemotherapy in Patients With Poor-Risk Rectal Cancer: the BRANCH Trial
Brief Title: Bevacizumab With Pelvic Radiotherapy And Primary Chemotherapy in Patients With Poor-Risk Rectal Cancer
Acronym: BRANCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANCH; 2008-003989-26 (EudraCT Number)
Record Dates: First submitted 2011-11-11; First posted 2011-11-29 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-09

CONDITIONS: Rectal Cancer
Keywords: locally advanced; high risk; preoperative therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Oxaliplatin; raltitrexed; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- preoperative chemoradiotherapy (Experimental): Preoperative radiation therapy and combination chemotherapy plus bevacizumab
  Interventions: Radiation: Radiation therapy; Drug: Oxaliplatin; Drug: Raltitrexed; Drug: levofolinic acid; Drug: 5-fluorouracil; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy will be administered at the total dose of 45 Gy, given with five weekly fractions over a period of 5 weeks. The daily fraction dose will be 1.8 Gy
Drug: Oxaliplatin — 100 mg/m2 on day 1 every 2 weeks for 3 cycles (for patients with resectable organ metastases (M1), an additional 2 cycles of chemotherapy will be given after radiation therapy)
Drug: Raltitrexed — 2.5 mg/m2 on day 1 every 2 weeks for 3 cycles (for patients with resectable organ metastases (M1) , an additional 2 cycles of chemotherapy will be given after radiation therapy)
Drug: levofolinic acid — 250 mg/m2 on day 2 every 2 weeks for 3 cycles (for patients with resectable organ metastases (M1), an additional 2 cycles of chemotherapy will be given after radiation therapy)
Drug: 5-fluorouracil — 800 mg/m2 on day 2 every 2 weeks for 3 cycles (for patients with resectable organ metastases (M1), an additional 2 cycles of chemotherapy will be given after radiation therapy)
Drug: Bevacizumab — will be given by intravenous infusion at the dose of 5 mg/kg concurrent with chemotherapy and radiotherapy every 2 weeks for 4 cycles from -14 days to start chemo-radiotherapy (classical schedule) or 4 days before the concurrent administration of chemotherapy and radiation therapy for 2 cycles if the number of TRG1 was not reached in the first stage (statistical design) with the classical schedule (for patients with resectable organ metastases (M1), one additional administration of bevacizumab will be given after radiation therapy)

SUMMARY:
The purpose of this study is to evaluate the use of chemotherapy, radiation therapy and bevacizumab before surgery in patients with locally advanced rectal cancer (LARC).

DETAILED DESCRIPTION:
To determine the pathological complete response (pCR-TRG1) rate in patients treated with 2 different schedule of bevacizumab plus primary chemotherapy and radiotherapy of the pelvic region when optimal surgery is applied.

Bevacizumab will be given by intravenous infusion at the dose of 5 mg/kg concurrent with chemotherapy and radiotherapy every 2 weeks for 4 cycles from -14 days to start chemo-radiotherapy (classical schedule) or 4 days before the concurrent administration of chemotherapy and radiation therapy for 2 cycles if the number of TRG1 was not reached in the first stage with the classical schedule Simon's methods will be used to calculate sample size.Setting a and b errors as 0.05 and 0.20, respectively, and defining as minimum activity of interest (p0) a TRG1 rate=30%. In order to demonstrate a TRG1 rate ≥50% (p1), at least 6 TRG1 on the first 15 patients, and at least 19 TRG1 on a total of 46 patients should be reported in the first and second stage, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of locally advanced rectal cancer (LARC) at high risk of recurrence (T4, N+, T3N0 with tumor located in the lower third of the rectum and/or circumferential resection margin (CRM) £5 mm), or LARC with resectable organ metastasis (M1).
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Life expectancy of at least 12 weeks
* Measurable and/or evaluable (resectable organ metastasis)lesions according to RECIST criteria
* Neutrophils > 1500 and Platelets > 100,000 /L
* Total bilirubin < or = 1.5 time the upper-normal limits (UNL) of the Institutional normal values and ASAT (SGOT) and/or ALAT (SGPT) < or = 2.5 x UNL, or < or = 5 x UNL in case of liver metastases, alkaline phosphatase < or = 2.5 x UNL, or < or = 5 x UNL in case of liver metastases.
* Creatinine clearance > 50 mL/min or serum creatinine < or = 1.5 x UNL
* Urine dipstick of proteinuria < 2+. Patients discovered to have > or = 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate < or = 1 g of protein/24 hr.
* Written informed consent.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating Center

Exclusion Criteria:

* Prior radiotherapy or chemotherapy for rectal cancer.
* Untreated brain metastases or spinal cord compression or primary brain tumours
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy or history of stroke).
* History of inflammatory bowel disease and/or acute/subacute bowel occlusion
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension
* Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes.
* Chronic, daily treatment with high-dose aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration.
* Treatment with any investigational drug within 30 days prior to enrolment.
* Patients with known allergy to Chinese hamster ovary cell proteins, or any of the components of the study medications
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal and squamous cell carcinoma or cervical cancer in situ
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, M.D., Principal Investigator — National Cancer Institute, Naples

RESULTS

PARTICIPANT FLOW:
Groups:
- Concomitant - Schedule A: Preoperative radiation therapy and combination chemotherapy plus bevacizumab
  Patients received three biweekly cycles of OXATOM/FUFA during RT. Bevacizumab was given 2 weeks before the start of chemoradiotherapy, and on the same day of chemotherapy for 3 cycles (concomitant-schedule A)
- Sequential - Schedule B: Preoperative radiation therapy and combination chemotherapy plus bevacizumab
  Patients received three biweekly cycles of OXATOM/FUFA during RT. Bevacizumab was given 4 days prior to the first and second cycle of chemotherapy (sequential-schedule B).
Period: Overall Study
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B
Started | 16 | 46
Completed | 11 | 40
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B | Total
Number analyzed (Participants) | 16 | 46 | 62
Age, Continuous [Median (Full Range); unit: years] | 55 [48 to 69] | 61 [43 to 74] | 58 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 25
  Male | 9 | 28 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Italian | 16 | 46 | 62
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 16 | 46 | 62
Distance of mesorectal Fascia (MRF) < 5 mm [Count of Participants; unit: Participants] | 13 | 35 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Tumor Regression Rate (TRG1)
Description: Complete tumor regression rate (TRG1) was the ratio of patients with TRG1, graded at surgical resection, and total patients included in the study, expressed in percentage.
  Tumor regression grade (TRG) was misured according to the Mandard Scale. Briefly,TRG1 was a complete tumor regression (regardless of the presence of acellular mucine lakes), and TRG2 was a nearly complete tumor regression with extensive fibrosis; TRG3 presented with clear evidence of residual cancer cells but with predominant fibrosis;TRG4 was a residual of cancer cells outgrowing fibrosis; TRG5 was the absence of regressive changes.
Time Frame: In 8 weeks after completion of chemoradiotherapy
Measure: Number; unit: percentage of participants
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B
Number analyzed (Participants) | 16 | 46
percentage of participants | 12.5 | 50

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Time Frame: Up to 8 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B
Number analyzed (Participants) | 16 | 46
Participants | 7 | 22

3. Secondary Outcome: Number of Patients With Sphincter Preservation
Description: Sphincter preservation in patients with tumor < 5 cm from anal verge in 8 weeks after chemoradiation therapy
Time Frame: In 8 weeks after chemoradiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B
Number analyzed (Participants) | 16 | 46
Participants | 13 | 41

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated from the date of the initial treatment until tumor progression or relapse, death for any cause or last follow up.
  Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 10 years
Population: PFS for the schedule A was not calculated because the number of TRG1 (2 out of 16 patients) was statistically inconsistent with the hypothesis of activity (30%) to be tested and, consequently, the accrual was early terminated.
Measure: Number; unit: participants
Arm/Group | Sequential - Schedule B | Concomitant - Schedule A
Number analyzed (Participants) | 46 | 16
participants | 37 | 11

5. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from the date of initial treatment to the date of death for any cause or last follow up.
Time Frame: 10 years
Population: OS for the schedule A was not calculated because the number of TRG1 (2 out of 16 patients) was statistically inconsistent with the hypothesis of activity (30%) to be tested and, consequently, the accrual was early terminated.
Measure: Number; unit: participants
Arm/Group | Sequential - Schedule B | Concomitant - Schedule A
Number analyzed (Participants) | 46 | 16
participants | 40 | 11

6. Secondary Outcome: Clinical Response Rate
Description: Clinical response was assessed before surgery with the same imaging modalities that were used for the inclusion in the study.
  Clinical response rate was the ratio between complete and partial response, evaluated by RECIST CRITERIA, and total of patients evaluated, expressed in percentage of patients.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 7 weeks after chemoradiation therapy up to 11 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Sequential - Schedule B | Concomitant - Schedule A
Number analyzed (Participants) | 46 | 16
percentage of participants | 40 | 20

7. Secondary Outcome: Patients With Metastatic Lymphnodes at Pathology Exam After Surgery
Description: Number of patients with metastatic lymphnodes at pathology exam after surgery.
Time Frame: In 8 weeks after chemoradiation therapy completion
Measure: Number; unit: participants
Arm/Group | Sequential - Schedule B | Concomitant - Schedule A
Number analyzed (Participants) | 46 | 16
participants | 14 | 5

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Concomitant - Schedule A | Sequential - Schedule B
All-Cause Mortality (participants affected / at risk) | 5/16 | 6/46
Serious Adverse Events (participants affected / at risk) | 7/16 | 14/46
Other Adverse Events (participants affected / at risk) | 7/16 | 22/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant - Schedule A (N=16) | Sequential - Schedule B (N=46)
Neutropenia (Blood and lymphatic system disorders) | 7 | 14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant - Schedule A (N=16) | Sequential - Schedule B (N=46)
Diarrhoea (Gastrointestinal disorders) | 6 | 16
Nausea/Vomiting (Gastrointestinal disorders) | 7 | 22
Proctitis (Gastrointestinal disorders) | 4 | 14
Asthenia (General disorders) | 4 | 10
Hypertension (Blood and lymphatic system disorders) | 4 | 11
Neutropenia (Blood and lymphatic system disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes